CLINICAL TRIAL: NCT05621421
Title: The Implementation of Intravascular Ultrasound and Fractional Flow Reserve in the Percutaneous Treatment of Very Long Coronary Artery Lesions
Status: Completed | Type: Observational
Sponsor: Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University (Other)
Responsible Party: Principal Investigator, Povilas Budrys, Principal investigator, Vilnius University Hospital Santaros Klinikos
Other Study IDs: 19-C-1252
Record Dates: First submitted 2022-11-03; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with long coronary artery lesions: Consecutive patients with functionally significant (FFR ≤ 0.8) long lesion requiring a stent length of ≥ 30mm to undergo FFR and IVUS guided PCI.
  Interventions: Procedure: FFR and IVUS guided PCI

INTERVENTIONS:
Procedure: FFR and IVUS guided PCI — PCI to the long lesion guided with FFR and IVUS

SUMMARY:
A single center, prospective, observational study to investigate the impact of intravascular ultrasound (IVUS) on the functional percutaneous coronary intervention (PCI) result (assessed with fractional flow reserve (FFR)) and one-year target vessel failure (TVF) rate after percutaneous treatment of long coronary artery lesions

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome (stable angina; staged PCI to other lesions after acute myocardial infarction with ST segment elevation);
* Acute coronary syndrome without ST segment elevation (unstable angina or myocardial infarction without ST segment elevation);
* Functionally significant (FFR ≤ 0.8) lesion requiring a stent length of ≥ 30 mm and amenable for percutaneous coronary intervention.

Exclusion Criteria:

* Patient's age ≤ 18 years;
* Acute myocardial infarction with ST segment elevation;
* Treatment with dual antiplatelet therapy contraindicated;
* Survival expectancy ≤ 1 year;
* Known allergy to sirolimus, everolimus or zotarolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with functionally significant long coronary artery lesions amenable to percutaenous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with optimal physiology result | 1 day
  Post PCI FFR value ≥ 0.9
The proportion of patients with optimal anatomy result | 1 day
  If all the four following IVUS criteria met: (1) good stent apposition; (2) good stent expansion (minimal stent area (MSA) >90% of distal reference lumen area and/or MSA ≥5.5mm2); (3) plaque burden 5mm proximal and distal to the stent <50%); (4) no stent edge dissection.
The proportion of patients with optimal physiology and anatomy result | 1 day
  Post PCI FFR value ≥ 0.9 and all four IVUS criteria met

SECONDARY OUTCOMES:
The rate of target vessel failure (TVF) | 12 months post PCI follow up
  Composite endpoint (target vessel related death (TV-death), target vessel related myocardial infarction (TV-MI), ischemia driven target vessel revascularization (TV-R))

CONTACTS AND LOCATIONS:
Overall Officials: Giedrius Davidavicius, PhD, Prof, Study Chair — Vilnius University Hospital Santaros Klinikos
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided